CLINICAL TRIAL: NCT02597023
Title: The Efficacy of Oral Mitoquinone (MitoQ) Supplementation for Improving Physiological in Middle-aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0402
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Aging
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MitoQ (Experimental): MitoQ, 20 mg per day for six weeks
  Interventions: Drug: MitoQ; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, inert excipient, one time per day for six weeks
  Interventions: Drug: MitoQ; Drug: Placebo

INTERVENTIONS:
Drug: MitoQ — Mitoquinone pill, 20 mg/day
  Other Names: mitoquinone
Drug: Placebo — Placebo pill with inert excipient, 1 time/day
  Other Names: placebo pill

SUMMARY:
The purpose of this study is to assess the efficacy of supplementation with the mitochondria-targeted antioxidant, mitoquinone (MitoQ), for improving physiological function (vascular, motor, and cognitive) in middle-aged and older adults.

DETAILED DESCRIPTION:
Overall, the proposed research project has the long-term potential to influence clinical practice by establishing novel therapies for treating multiple domains of age-associated physiological dysfunction and thereby reducing the risk of clinical disease and disability.

ELIGIBILITY:
Inclusion Criteria:

* Women will be confirmed as postmenopausal (either natural or surgical) based on cessation of menses for >1 year.
* Ability to provide informed consent
* Baseline brachial flow-mediated dilation (FMD) < 6%Δ (rationale: non-invasive screening to ensure exclusion of subjects with exceptionally high baseline endothelial function.
* Ability to perform motor and cognitive tests (e.g., can rise from a chair, walk for 2 min, climb 10 stairs)
* Willing to accept random assignment to condition

Exclusion Criteria:

* Current smoking
* Having past or present alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders
* Body mass index (BMI) >40 kg/m2 (FMD measurements can be inaccurate in severely obese patients)
* Chronic clinical diseases (e.g., coronary artery/peripheral artery/cerebrovascular diseases, diabetes, chronic kidney disease requiring dialysis, neurological disorders or diseases that may affect motor/cognitive functions [multiple sclerosis, Parkinson's disease, polio, Alzheimer's disease, dementia or other brain diseases of aging]), except hypertension and hyperlipidemia
* Regular vigorous aerobic/endurance exercise (>3 vigorous bouts/week).
* Not weight stable in the prior 3 months (>2 kg weight change) or unwilling to remain weight stable throughout study (rationale: recent weight change or weight loss can influence vascular function.
* Current treatment or recent cessation (< 3 mo) of hormone replacement therapy
* Moderate or severe peripheral artery disease (ankle-brachial index <0.7).
* A graded exercise test will be performed by all subjects, if there is physician concern or an adverse event, the subject will not participate in a maximal oxygen consumption (VO2max) test (this will be determined in accordance with stated contraindications for exercise testing provided by the American Heart Association).
* Thyroid disease that is not controlled by medications or <3 month's use of a particular medication and/or dosage (uncontrolled thyroid diseases are associated with alterations in vascular function).

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent dilation | 6 weeks
  Flow-mediated dilation

SECONDARY OUTCOMES:
Systemic markers of oxidative stress | 6 weeks
  Oxidized LDL levels in blood.
Motor function | 6 weeks
  NIH Toolbox motor test battery
Cognitive function | 6 weeks
  NIH Toolbox cognition test battery
Arterial Stiffness | 6 weeks
  Aortic pulse wave velocity
Endothelial cell markers of oxidative stress | 6 weeks
  Nitrotyrosine levels in biopsied endothelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Rossman, PhD, Study Director — University of Colorado, Boulder; Douglas R Seals, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Clinical Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- [Derived] Rossman MJ, Santos-Parker JR, Steward CAC, Bispham NZ, Cuevas LM, Rosenberg HL, Woodward KA, Chonchol M, Gioscia-Ryan RA, Murphy MP, Seals DR. Chronic Supplementation With a Mitochondrial Antioxidant (MitoQ) Improves Vascular Function in Healthy Older Adults. Hypertension. 2018 Jun;71(6):1056-1063. doi: 10.1161/HYPERTENSIONAHA.117.10787. Epub 2018 Apr 16. PMID 29661838
- See also: Description of our Research Laboratory — http://www.colorado.edu/intphys/research/cardiovascular.html